CLINICAL TRIAL: NCT06115577
Title: Receptivity of Endometrial Tissue and Peripheral Blood Mononuclear Cells in the Pathogenetic Rationale for the Management of Postmenopause Patients With Endometrial Proliferative Processes
Brief Title: Endometrial Tissues and Mononuclear Cells Receptivity in Pathogenesis of Endometrial Proliferative Processes
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 210
Record Dates: First submitted 2023-10-24; First posted 2023-11-03 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: Endometrial Hyperplasia Without Atypia; Endometrial Hyperplasia With Atypia; Endometrial Cancer; Peripheral Blood Mononuclear Cells; Postmenopause; Estrogen Receptor; Progesterone Receptor
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- endometrial polyp: pathology according to histological examination
  Interventions: Diagnostic Test: endometrial tissue and peripheral blood mononuclear cells receptivity
- endometrial hyperplasia without atypia: pathology according to histological examination
  Interventions: Diagnostic Test: endometrial tissue and peripheral blood mononuclear cells receptivity
- atypical endometrial hyperplasia: pathology according to histological examination
  Interventions: Diagnostic Test: endometrial tissue and peripheral blood mononuclear cells receptivity
- endometrial cancer: pathology according to histological examination
  Interventions: Diagnostic Test: endometrial tissue and peripheral blood mononuclear cells receptivity

INTERVENTIONS:
Diagnostic Test: endometrial tissue and peripheral blood mononuclear cells receptivity — Participants investigated the expression level of estrogen and progesterone receptors (ERα, ERβ, GPER, PRA, PRB, mPR, PGRmC1) by RT-PCR in pathological endometrial tissue and peripheral blood mononuclear cells. GABDH was used as a comparison gene.

SUMMARY:
A prospective observational study of endometrial tissue and peripheral blood mononuclear cells receptivity to sex steroid hormones in postmenopausal patients with endometrial proliferative processes

DETAILED DESCRIPTION:
Endometrial cancer is in third place among cancer diseases in female population of Russia. The peak morbidity occurs during the postmenopausal period. In this regard, early diagnosis of previous endometrial proliferative processes and effective methods for their treatment are relevant. However, failures with hormonal therapy are often observed. This may be due to the low receptivity of the pathological tissue. It is also known that the functional activity of immunocompetent cells is controlled by the immune system, however, studies of the receptivity of peripheral blood mononuclear cells to sex steroid hormones were carried out in healthy blood donors. Changes in mononuclear cells receptivity may be one of the pathogenetic links in the development of endometrial proliferative processes and endometrial cancer. This may also influence the effectiveness of their treatment. In this regard, the purpose of the study is to evaluate the role of the expression of estradiol and progesterone receptor genes in endometrial tissue and peripheral blood mononuclear cells in the occurrence of endometrial proliferative processes in postmenopausal patients with a pathogenetic justification for the choice of treatment method. To achieve this goal, the investigators investigated the expression level of estrogen and progesterone receptors (ERa, ERb, GPER, PRA, PRB, mPR, PGRmC1) by RT-PCR in pathological endometrial tissue and peripheral blood mononuclear cells. GABDH was used as a comparison gene. The data obtained made it possible to determine the significance of mononuclear cell receptivity in the pathogenesis of endometrial proliferative processes.

ELIGIBILITY:
Inclusion Criteria:

* endometrial polyps
* endometrial hyperplasia
* atypical endometrial hyperplasia
* endometrial cancer

Exclusion Criteria:

* hormonal treatment (estrogen-progestogens, gestagens, gonadotropin-releasing hormone agonists, menopausal hormone therapy and tamoxifen) for 6 months before the study
* uterine fibroids, larger than 6-7 pregnancy weeks
* pathology of the uterine appendages according to ultrasound pelvis
* inflammatory diseases of various localization at the time of taking the material

Ages: 53 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included 92 patients with endometrial proliferative processes: endometrial polyp - 37, endometrial hyperplasia without atypia - 7, atypical endometrial hyperplasia - 8, endometrial cancer - 40
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
endometrial tissue and peripheral blood mononuclear cells receptivity | through study completion, an average of 1 year
  Expression level of ERα, ERβ, GPER, PRA, PRB, mPR, PGRmC1 in endometrial tissue and peripheral blood mononuclear cells in patients with endometrial polyps, endometrial hyperplasia, atypical endometrial hyperplasia, endometrial cancer

CONTACTS AND LOCATIONS:
Overall Officials: Dina Gutorova, PhD, Principal Investigator — Pirogov Russian National Research Medical University

DOCUMENTS (1):
  • Study Protocol (2012-10-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT06115577/Prot_000.pdf